CLINICAL TRIAL: NCT05538429
Title: Comparison of Analgesic Effect and Postoperative Recovery of Serratus Anterior Plane Block Combined With Erector Spinae Plane Block and Thoracic Paravertebral Block After Thoracoscopic Surgery
Brief Title: Comparison of Analgesic Effect and Postoperative Recovery of SAPB Combined With ESPB and TPB After Thoracoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhangyi (Other)
Responsible Party: Sponsor-Investigator, Zhangyi, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 1000012129
Record Dates: First submitted 2022-01-27; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Thoracoscopic Surgery; Nerve Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB&SAPB (Experimental): erector spinal plane block combined with serratus anterior plane block
  Interventions: Procedure: erector spinal plane combined with serratus anterior plane block
- TPVB (Active Comparator): thoracic paravertebral block
  Interventions: Procedure: erector spinal plane combined with serratus anterior plane block

INTERVENTIONS:
Procedure: erector spinal plane combined with serratus anterior plane block — The experimental group received ultrasound-guided erector spinal block combined with serratus anterior plane block, and erector spinal block was performed at the T5 and T7 levels with 10ml 0.4% ropivacaine for each level, and 20ml 0.4% ropivacaine for serratus anterior plane block. The control group received ultrasound-guided thoracic paravertebral block at T5 and T7 levels, respectively, with 20ml 0.4% ropivacaine at each level.
  Other Names: thoracic paravertebral block

SUMMARY:
After thoracoscopic surgery, patients still face moderate to severe pain. How to effectively control pain and promote postoperative recovery of patients is a challenging problem. Thoracic paraspinal block is effective in controlling pain after thoracoscopic surgery, but it also carries the risk of difficulty in operation and puncture of the pleura. In recent years, erector spinal plane block and serratus anterior plane block have been used for postoperative analgesia after thoracoscopic surgery. The purpose of this study was to explore whether erector spinal plane combined with serratus anterior plane block can replace thoracic paravertebral block and provide a more complete analgesia after thoracoscopic surgery. Therefore, this study is of great clinical significance.

DETAILED DESCRIPTION:
In a double-blind randomized controlled study, investigators allocated 92 patients undergoing VATS to either SAPB Combined With ESPB or TPB, with both groups receiving otherwise standardized treatment, including multimodal analgesia. The primary outcome was 24-hr opioid consumption. Secondary outcomes included the number of survival analgesia at 1, 2, 4, 8, and 24 hours postoperatively ,VAS scores was assessed during resting and coughing statuses at 1, 2, 4, 8, and 24 hours postoperatively, pulmonary function indexes before and 1, 4, 24 hours after surgery , QOR-15 scores before and 24 hours after surgery, postoperative complications and recovery time nodes drainage tube removal time, discharge time.

ELIGIBILITY:
Inclusion Criteria:

1. American ASA Grade I-III;
2. Age: 18 ~ 70 years old;

3 BMI 19 ~ 28kg/m2;

4. Patients with elective thoracoscopic partial pneumonectomy under general anesthesia;

5 Informed Consent has been signed.

Exclusion Criteria:

1. Use opioid analgesics on a daily basis or have a history of opioid abuse;
2. History of ipsilateral thoracotomy;
3. Allergic to any of the drugs used in the study, or have a history of drug allergy;
4. Mental or nervous system diseases, motor or sensory deficits;

5 there is coagulation dysfunction;

6. Cognitive dysfunction, unable to cooperate with research;

7. Severe renal, hepatic or cardiac dysfunction;

8. Chest wall and spine trauma, infection, deformity and other cases where nerve block cannot be performed;

9. Participated in other clinical trials within the 3 months prior to study inclusion;

10. Investigators consider other reasons unsuitable for clinical trial participants;

11. Patients refuse to participate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
The dose of opioids used | 24 hours after surgery
  dosage of analgesic pump

SECONDARY OUTCOMES:
The dose of opioids used | 1hour, 2hours, 4hours, 8hours and 48hours postoperatively after surgery
  dosage of analgesic pump
The number of survival analgesia | 1hour, 2hours, 4hours, 8hours, 24hours and 48hours after surgery
  times of rescue analgesia
VAS scores at resting and coughing state | 1hour, 2hours, 4hours, 8hours, 24hours and 48hours after surgery
  visual analog pain scale
pulmonary function indexes | Preoperative, postoperative 1hour, postoperative 4hours and postoperative 24hours
  FVC (L)
QOR-15 scores | before and 24 hours after surgery
  The highest score is 150,the lowest score is 0. The higher the score, the better off the patient was.
Postoperative complications and recovery time nodes | follow up patients for an average of half a month
  drainage tube removal time, length of stay, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology., Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/29/NCT05538429/Prot_SAP_ICF_000.pdf